CLINICAL TRIAL: NCT06944210
Title: Evaluation of the Antioxidant and Anti-Inflammatory Capacities of the 'Rosy Red Valencia' and 'Olinda Valencia' Sweet Orange Varieties in Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22923441
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Oranges; Lycopene; Healthy; Oxidative stress; Inflammation; gene expression
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Rosy Red Valencia' sweet orange variety (Experimental): The participants of this group consume 'Rosy Red Valencia' sweet oranges
  Interventions: Other: 'Rosy Red Valencia' sweet orange
- 'Olinda Valencia' sweet orange variety (Experimental): The participants of this group consume 'Olinda Valencia' sweet oranges
  Interventions: Other: 'Olinda Valencia' sweet oranges

INTERVENTIONS:
Other: 'Rosy Red Valencia' sweet orange — The participants consume 2 'Rosy Red Valencia' sweet oranges daily for 4 weeks
  Arms: 'Rosy Red Valencia' sweet orange variety
Other: 'Olinda Valencia' sweet oranges — The participants consume 2 'Olinda Valencia' sweet oranges daily for 4 weeks
  Arms: 'Olinda Valencia' sweet orange variety

SUMMARY:
This study aims to evaluate the antioxidant and anti-inflammatory effects of acute and chronic consumption of two sweet orange (Citrus sinensis) varieties-'Rosy Red Valencia', which is rich in carotenoids such as lycopene, phytoene, and phytofluene, and 'Olinda Valencia', which lacks these carotenoids-in healthy adults. In this 4-week, randomized, parallel-arm clinical trial, participants will consume either 'Rosy Red Valencia' or 'Olinda Valencia' oranges daily. The study will assess the effects of sweet orange intake on markers of oxidative stress and inflammation, plasma carotenoid concentrations, gene expression in peripheral blood mononuclear cells, and gut health. Findings from this study may help identify potential health benefits associated with specific carotenoid profiles in sweet oranges and provide insights into their role in modulating inflammation and oxidative stress.

DETAILED DESCRIPTION:
The health benefits of orange consumption have been described; however, the specific bioactive compounds responsible for these effects, as well as the underlying mechanisms of action, are not fully understood. There are several varieties of sweet oranges, each with a unique phytochemical profile and potentially distinct health-promoting properties. The 'Rosy Red Valencia' sweet orange is enriched in carotenoids such as lycopene, phytoene, and phytofluene, whereas the commonly consumed 'Olinda Valencia' contains negligible levels of these compounds.

This randomized, parallel-arm clinical trial aims to evaluate and compare the antioxidant and anti-inflammatory effects of 'Rosy Red Valencia' and 'Olinda Valencia' sweet orange consumption in healthy men and women. Participants will be randomized to consume one of the two orange varieties twice daily for four weeks.

The study includes both an acute phase (1-day consumption) and a chronic phase (4-week daily consumption). Blood samples will be collected at baseline, after 1 day, and after 4 weeks of consumption to assess changes in plasma carotenoid concentrations, markers of oxidative stress and inflammation, and gene expression profiles in peripheral blood mononuclear cells. Fecal samples will be collected at baseline and after 4 weeks to assess the effects on gut microbiota composition. By evaluating and comparing the biological effects of these two orange varieties, the study aims to elucidate the role of specific carotenoids in mediating the health benefits of sweet orange consumption.

ELIGIBILITY:
Inclusion Criteria

* Healthy men and women
* Age Range: 25-40 years
* Body mass index (BMI) with values between 21 and 29.9 kg^m2
* Willingness to accept randomization, undergo the testing and intervention procedures, and deliver blood and stool samples
* Willingness to refrain from consuming foods rich in lycopene, phytoene, and phytofluene and limit the intake of some polyphenol-rich foods
* Willingness to discontinue the use of antioxidant supplements (such as carotenoid, polyphenol supplements), prebiotics and/or probiotics

Exclusion Criteria:

* Pregnancy/lactation
* History of cardiovascular diseases, diabetes, uncontrolled hypertension, heart failure, stroke, liver, gallbladder, kidney, thyroid disease, gastrointestinal, autoimmune disorder, or cancer.
* Psychiatric disease that interferes with the understanding and implementation of the intervention
* History of eating disorders (such as bulimia nervosa and anorexia nervosa) in the last 5 years
* Current smokers
* Vegan, vegetarian, or other special diets (e.g., keto, paleo)
* Use of antibiotics or laxatives in the previous month
* History of substance abuse or alcohol abuse
* involvement in a weight loss intervention program within the past month or weight change > 10%
* Self-report of allergic reactions to study products or their phytochemicals.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-17 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Levels of lycopene and noncolored carotenoids | 0, 1 day, 4 weeks
  Levels in plasma

SECONDARY OUTCOMES:
Oxidative stress markers | 0, 1 day, 4 weeks
  Markers of oxidative stress in plasma/ blood cells
Inflammatory markers | 0, 1 day, 4 weeks
  Markers of inflammation in plasma
Gene expression | 0, 1 day, 4 weeks
  Gene expression in Peripheral Blood Mononuclear Cells (PBMCs)
Lipid/metabolic profile | 0, 4 weeks
  Measured in blood samples
Blood pressure | 0, 4 weeks
Microbiota composition | 0, 4 weeks
  From stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo G Macknezie, PhD, Study Director — Univeristy of California Davis
Locations (1):
- Nutrition Department, Ragle Facility, University of California Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No